CLINICAL TRIAL: NCT00002894
Title: A RANDOMISED TRIAL OF PACLITAXEL (TAXOL) IN COMBINATION WITH PLATINUM CHEMOTHERAPY VS. CONVENTIONAL PLATINUM-BASED CHEMOTHERAPY IN THE TREATMENT OF WOMEN WITH RELAPSED OVARIAN CANCER
Brief Title: Platinum-based Chemotherapy With or Without Paclitaxel in Treating Patients With Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065217; MRC-ICON4; EU-96051; ISRCTN47434271
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2001-02

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Cisplatin; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of platinum-based chemotherapy with or without paclitaxel in treating patients with relapsed ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare survival of patients with relapsed ovarian epithelial or peritoneal cancer treated with paclitaxel and either carboplatin or cisplatin vs conventional platinum-based chemotherapy.
* Compare the quality of life and health economics of these regimens in these patients.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive platinum-based chemotherapy (that is familiar to the oncologist and used routinely by the center) comprising either cisplatin or carboplatin alone or cisplatin in combination with other drugs.
* Arm II: Patients receive paclitaxel IV over 3 hours followed by either carboplatin or cisplatin.

Treatment for both arms continues every 3 weeks for up to 6 courses in the absence of unacceptable toxicity.

Quality of life is assessed.

Patients are followed at 6 months, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 800 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Ovarian epithelial cancer or serous peritoneal carcinoma that has relapsed after prior chemotherapy

  * Progression-free interval (from end of last treatment) of at least 6 months
* Measurable disease not required

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2 times normal

Renal:

* Not specified

Other:

* No sepsis
* No contraindication to chemotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 1996-03; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A. Ledermann, MD, Study Chair — University College London Hospitals
Locations (1):
- Middlesex Hospital- Meyerstein Institute, London, England, United Kingdom

REFERENCES:
- [Background] Kushner DM, Connor JP, Sanchez F, Volk M, Schink JC, Bailey HH, Harris LS, Stewart SL, Fine J, Hartenbach EM; Wisconsin Oncology Network. Weekly docetaxel and carboplatin for recurrent ovarian and peritoneal cancer: a phase II trial. Gynecol Oncol. 2007 May;105(2):358-64. doi: 10.1016/j.ygyno.2006.12.018. Epub 2007 Jan 29. PMID 17258800
- [Background] Pfisterer J, Ledermann JA. Management of platinum-sensitive recurrent ovarian cancer. Semin Oncol. 2006 Apr;33(2 Suppl 6):S12-6. doi: 10.1053/j.seminoncol.2006.03.012. PMID 16716798
- [Result] Ledermann JA: Randomised trial of paclitaxel in combination with platinum chemotherapy versus platinum-based chemotherapy in the treatment of relapsed ovarian cancer (ICON4/OVAR2.2). [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1794, 446, 2003.
- [Result] Parmar MK, Ledermann JA, Colombo N, du Bois A, Delaloye JF, Kristensen GB, Wheeler S, Swart AM, Qian W, Torri V, Floriani I, Jayson G, Lamont A, Trope C; ICON and AGO Collaborators. Paclitaxel plus platinum-based chemotherapy versus conventional platinum-based chemotherapy in women with relapsed ovarian cancer: the ICON4/AGO-OVAR-2.2 trial. Lancet. 2003 Jun 21;361(9375):2099-106. doi: 10.1016/s0140-6736(03)13718-x. PMID 12826431